CLINICAL TRIAL: NCT05155566
Title: Treatment Patterns And Clinical Outcomes Among Patients in Latin America Receiving First Line Palbociclib Combinations For HORMONE RECEPTOR POSITIVE/ HUMAN EPIDERMAL GROWTH FACTOR RECEPTOR 2 NEGATIVE (HR+/HER2-) Advanced/Metastatic Breast Cancer In Real World Settings
Brief Title: Treatment Patterns And Clinical Outcomes Among Patients in Latin America Receiving First Line Palbociclib Combinations For HR+/HER2- Advanced/Metastatic Breast Cancer In Real World Settings.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481125; IRIS LATAM (Other: Alias Study Number)
Record Dates: First submitted 2021-12-09; First posted 2021-12-13 (Actual); Results first posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer Metastatic
Keywords: human epidermal growth factor receptor 2 negative (HER2-); hormone receptor positive (HR+); advanced breast cancer (ABC); metastatic breast cancer (MBC)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Breast Cancer Patients: HR + /HER2- Advanced/Metastatic Breast Cancer patients in Latin America

SUMMARY:
To describe patient demographics, clinical characteristics, treatment patterns and clinical outcomes of adult female patients who have received palbociclib combination treatments as first line therapy, regardless of combination partner and labelled use in real world settings across Latin America.

ELIGIBILITY:
Physician inclusion criteria:

* Oncologist or gynecologist.
* Responsible for treating ≥4-10 (depending on country) ABC/MBC patients who meet the eligibility criteria.
* Agrees to participate in the study and complete the case report forms (CRFs) within the data collection period.

Patient inclusion criteria:

* HR+/HER2- breast cancer diagnosis with confirmed metastatic or advanced disease.
* Received palbociclib as a first line therapy.
* No prior or current enrolment in an interventional clinical trial for ABC/MBC.
* Minimum of six months of follow up data since palbociclib initiation.

Physician exclusion criteria:

* Qualified less than 2 years ago or more than 35 years ago.
* Participated in observational research for ABC/MBC in the last 3 months.
* Have not prescribed either palbociclib plus fulvestrant or palbociclib plus aromatase inhibitor as first line therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective medical data review of patients who have received palbociclib combination treatments as first line treatment regardless of combination partner and labelled use in Argentina, Chile, Peru, Mexico and a combined sample in Costa Rica and Panama.
Sampling Method: Non-Probability Sample
Enrollment: 847 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer country office, Buenos Aires, Argentina
- Adelphi Mill, Bollington, Cheshire, SK10 5JB, UK, Bollington, Chesshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481125

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with hormone receptor (HR) positive/Human Epidermal Growth Factor Receptor 2 (HER2) negative advanced or metastatic breast cancer who received palbociclib in combination with aromatase inhibitor or fulvestrant as first-line therapy were observed. Data was collected retrospectively from participants medical records and evaluated over approximately 22 months of this study.
Groups:
- Palbociclib + Aromatase Inhibitor: Participants with HR positive/HER2 negative advanced or metastatic breast cancer who received palbociclib as a first-line therapy along with aromatase inhibitor were observed during this retrospective study.
- Palbociclib + Fulvestrant: Participants with HR positive/HER2 negative advanced or metastatic breast cancer who received palbociclib as a first-line therapy along with fulvestrant were observed during this retrospective study.
Period: Overall Study
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Started | 574 | 273
Completed | 574 | 273
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) comprised of participants for whom a complete medical record review was conducted.
Groups:
- Total: Total of all reporting groups
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant | Total
Number analyzed (Participants) | 574 | 273 | 847
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (11.4) | 58.3 (10.2) | 60.0 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 574 | 273 | 847
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 1 | 0 | 1
  Native American | 5 | 3 | 8
  Asian-Indian subcontinent | 1 | 0 | 1
  Asian - other | 0 | 1 | 1
  Chinese | 0 | 1 | 1
  Hispanic/Latino | 348 | 180 | 528
  Middle Eastern | 1 | 0 | 1
  Mixed race | 31 | 9 | 40
  White/Caucasian | 175 | 61 | 236
  Afro-Caribbean | 3 | 6 | 9
  Other | 7 | 4 | 11
  Black | 0 | 3 | 3
  Prefer not to answer | 2 | 5 | 7
Number of Participants According to Menopause Status at Palbociclib Initiation [Count of Participants; unit: Participants] — Menopause status at palbociclib initiation including menopause induced by Luteinizing hormone-releasing hormone (LHRH) suppression, menopause induced by surgery, natural menopause, perimenopausal and premenopausal were reported.
  Participants
    Menopause Induced by LHRH Suppression | 33 | 15 | 48
    Menopause Induced by Surgery | 49 | 10 | 59
    Natural Menopause | 483 | 234 | 717
    Perimenopausal | 2 | 12 | 14
    Premenopausal | 7 | 2 | 9
Number of Participants According to Type of Insurance Plan [Count of Participants; unit: Participants] — Number of participants according to the type of insurance plan was reported
  Participants
    Argentina-Servicio de Salud Publico | 51 | 5 | 56
    Argentina-Seguridad Social | 176 | 58 | 234
    Argentina-PrivadoPrepagas | 123 | 56 | 179
    Mexico-ISSSTE | 7 | 0 | 7
    Mexico-Sedena | 0 | 1 | 1
    Mexico- PEMEX | 4 | 3 | 7
    Mexico-Aseguradora privada | 53 | 6 | 59
    Mexico-IMSS | 10 | 4 | 14
    Mexico-SSA | 5 | 0 | 5
    Mexico-Aseguradoras privadas | 24 | 6 | 30
    Chile-FONASA (El Fondo Nacional de Salud) | 1 | 5 | 6
    Chile-ISAPRE (Instituciones de Salud Previsional) | 2 | 0 | 2
    Costa rica/Panama-CSS (Caja de seguridad social) | 28 | 8 | 36
    Costa rica/Panama-Aseguradora privada | 5 | 0 | 5
    Colombia-Contributive regime (POS-C) | 57 | 82 | 139
    Colombia-Subsidized regime (POS-S) | 22 | 16 | 38
    Colombia-Special regime (i.e. teacher or military) | 1 | 22 | 23
    Colombia-Unknown | 5 | 1 | 6
Number of Participants With Positive Biomarker Status [Count of Participants; unit: Participants] — Number of participants with positive status for following biomarkers: breast cancer type 1 (BRCA1) gene, breast cancer type 2 (BRCA2), androgen receptor and estrogen receptor 1 (ESR1) mutation were reported.
  Participants
    BRCA1 | 11 | 59 | 70
    BRCA2 | 5 | 58 | 63
    Androgen receptor | 31 | 71 | 102
    ESR1 mutation | 0 | 36 | 36
Number of Participants According to Family History of Breast Cancer [Count of Participants; unit: Participants] — Number of participants according to their family history of breast cancer as yes, no and unknown were reported.
  Participants
    Yes | 115 | 57 | 172
    No | 421 | 193 | 614
    Unknown | 38 | 23 | 61
Number of Participants According to Stage of Initial Breast Cancer [Count of Participants; unit: Participants] — Number of participants according to stage at initial breast cancer diagnosis is presented. Staging used was American Joint Committee on Cancer (AJCC) Tumor Node Metastasis (TNM), where Stage 0=noninvasive ductal carcinoma in situ; Stage 1= tumor size up to 2 centimeters (cm) and no lymph node involved; Stage 2= tumor size between 2 to 5 cm, cancer has spread to lymph nodes; Stage 3a= any size tumor, spread to 4 to 9 lymph nodes.; Stage 3b=tumor has spread to chest wall; Stage 3c= any size tumor, spread to 10 or more lymph nodes; Stage 4 (metastatic)= any size tumor has spread to other organs.
  Participants
    Stage 0 | 0 | 1 | 1
    Stage 1 | 21 | 11 | 32
    Stage 2 | 111 | 91 | 202
    Stage 3a | 86 | 144 | 230
    Stage 3b | 41 | 5 | 46
    Stage 3c | 21 | 1 | 22
    Stage 4 | 294 | 20 | 314
Number of Participants With Metastases to Lymph Nodes [Count of Participants; unit: Participants] — Number of participants with metastases to lymph nodes (regional and distal) were presented. Population: Here, number anaylzed signifies participants evaluable for this baseline measure.
  Participants
    Lymph nodes, Regional: number analyzed (Participants) | 485 | 203 | 688
    Lymph nodes, Regional | 85 | 12 | 97
    Lymph nodes, Distal: number analyzed (Participants) | 485 | 203 | 688
    Lymph nodes, Distal | 59 | 31 | 90
Number of Participants According to Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance status is used to measure quality of life of participants with grades ranging from 0 to 5; where Grade 0: Fully active; Grade 1: Restricted in physically strenuous activity but ambulatory; Grade 2: Ambulatory and capable of all self-care but unable to carry out any work activities; Grade 3: Capable of only limited self-care; Grade 4:Completely disabled and Grade 5: Dead. Higher scores indicated worsening of quality of life. Number of participants according to ECOG status were presented.
  Participants
    Grade 0 | 154 | 59 | 213
    Grade 1 | 307 | 110 | 417
    Grade 2 | 103 | 43 | 146
    Grade 3 | 6 | 32 | 38
    Grade 4 | 3 | 28 | 31
    Unknown | 1 | 1 | 2
Number of Participants According to Diagnosis for Which Palbociclib Combination was Prescribed [Count of Participants; unit: Participants] — Number of participants prescribed palbociclib combination treatment for advanced/metastatic breast cancer were presented.
  Participants | 574 | 273 | 847
Number of Participants According to Different Sites of Metastases [Count of Participants; unit: Participants] — Number of participants according to the sites of metastases was presented. Participant could have more than one site of metastases. Population: Here, number anaylzed signifies participants evaluable for this baseline measure.
  Participants
    Bone: number analyzed (Participants) | 485 | 203 | 688
    Bone | 374 | 140 | 514
    Lymph node: number analyzed (Participants) | 485 | 203 | 688
    Lymph node | 145 | 43 | 188
    Lung: number analyzed (Participants) | 485 | 203 | 688
    Lung | 156 | 54 | 210
    Liver: number analyzed (Participants) | 485 | 203 | 688
    Liver | 89 | 32 | 121
    Brain: number analyzed (Participants) | 485 | 203 | 688
    Brain | 8 | 2 | 10
    Skin/soft tissue: number analyzed (Participants) | 485 | 203 | 688
    Skin/soft tissue | 87 | 40 | 127
    Ovary: number analyzed (Participants) | 485 | 203 | 688
    Ovary | 3 | 6 | 9
    Other: number analyzed (Participants) | 485 | 203 | 688
    Other | 4 | 3 | 7
    Visceral disease: number analyzed (Participants) | 485 | 203 | 688
    Visceral disease | 221 | 84 | 305
    Non-visceral disease: number analyzed (Participants) | 485 | 203 | 688
    Non-visceral disease | 264 | 119 | 383
Number of Participants With De novo and Recurrent Breast Cancer [Count of Participants; unit: Participants] — Number of participants with de novo and recurrent breast cancer occurrence were reported
  Participants
    De Novo | 356 | 26 | 382
    Recurrent | 218 | 247 | 465
Number of Participants With Comorbidities Diagnosed in 12 Months Prior to Palbociclib Initiation [Count of Participants; unit: Participants] — Participants with their comorbidities diagnosed within 12 months prior to palbociclib initiation were reported. Population: Here, number anaylzed signifies participants evaluable for this baseline measure.
  Participants
    Bradyarrhythmias | 1 | 2 | 3
    Cerebrovascular disease | 7 | 3 | 10
    Congestive heart failure | 5 | 8 | 13
    Chronic pulmonary disease | 12 | 11 | 23
    Connective tissue disease | 1 | 0 | 1
    Dementia | 5 | 2 | 7
    Diabetes with end organ damage | 12 | 1 | 13
    Diabetes without end organ damage | 89 | 46 | 135
    Depression | 50 | 35 | 85
    Electrolyte abnormalities | 2 | 0 | 2
    Hypertension | 227 | 94 | 321
    Long QT syndrome | 1 | 0 | 1
    Mild liver disease | 7 | 8 | 15
    Moderate to severe renal disease | 5 | 23 | 28
    Myelosuppression | 2 | 0 | 2
    Myocardial infarction | 1 | 1 | 2
    Peptic ulcer disease | 18 | 9 | 27
    Peripheral vascular disease | 14 | 3 | 17
    Unstable angina | 2 | 2 | 4
    Unknown | 9 | 4 | 13
    Other | 21 | 9 | 30
    None | 257 | 106 | 363
Number of Participants Prescribed Palbociclib (Aromatase Inhibitor or Fulvestrant at First Line) [Count of Participants; unit: Participants] | 574 | 273 | 847
Age at Initial Breast Cancer Diagnosis [Mean (Standard Deviation); unit: Years] — Population: Here, number anaylzed signifies participants evaluable for this baseline measure.
  Years
    number analyzed (Participants) | 541 | 255 | 796
    (all) | 58.1 (12.0) | 55.2 (10.0) | 57.2 (11.5)
Age at Advanced Breast Cancer (ABC)/Metastatic Breast Cancer (mBC) Diagnosis [Mean (Standard Deviation); unit: Years] — Population: Here, number anaylzed signifies participants evaluable for this baseline measure.
  Years
    number analyzed (Participants) | 539 | 258 | 797
    (all) | 60.4 (11.7) | 58.3 (10.0) | 59.7 (11.2)
Time From Initial Breast Cancer Diagnosis to ABC/mBC Diagnosis [Median (Full Range); unit: Months] — Population: Here, number anaylzed signifies participants evaluable for this baseline measure.
  Months
    number analyzed (Participants) | 207 | 227 | 434
    (all) | 58.0 [0.0 to 397.5] | 25.1 [0.0 to 246.7] | 39.2 [0.0 to 397.5]
Time from ABC/mBC Diagnosis to Palbociclib Initiation [Median (Full Range); unit: Months] — The date of palbociclib treatment initiation was the study baseline. Here, time from ABC/mBC diagnosis to palbociclib initiation was reported. Population: Here, number anaylzed signifies participants evaluable for this baseline measure.
  Months
    number analyzed (Participants) | 539 | 258 | 797
    (all) | 1.8 [0.0 to 232.6] | 1.4 [0.0 to 128.1] | 1.7 [0.0 to 232.6]
Number of Participants With Adjuvant Treatments Received Since Breast Cancer Diagnosis [Count of Participants; unit: Participants] — Number of participants who received adjuvant chemotherapy and adjuvant endocrine therapy for early breast cancer treatment were reported.
  Participants
    Adjuvant Chemotherapy | 130 | 138 | 268
    Adjuvant endocrine therapy | 178 | 245 | 423
Number of Participants who Received Radiotherapy or Surgery [Count of Participants; unit: Participants] — Number of participants who received radiotherapy and surgery for early breast cancer were reported.
  Participants
    Radiotherapy | 177 | 200 | 377
    Surgery | 190 | 195 | 385
Duration of adjuvant endocrine therapy [Mean (Standard Deviation); unit: Months] — Duration of adjuvant endocrine therapy for early breast cancer treatment is presented. Population: Here, number anaylzed signifies participants evaluable for this baseline measure.
  Months
    number analyzed (Participants) | 178 | 245 | 423
    (all) | 40.7 (25.4) | 24.3 (22.4) | 31.2 (25.0)
Time Since end of Adjuvant Treatment [Median (Full Range); unit: Months] — Population: Data was not collected for this baseline measure
Time From Regimen Completion of Adjuvant Therapy to Diagnosis of ABC/mBC [Median (Full Range); unit: Months] — Population: Data was not collected for this baseline measure
Time From Initial Breast Cancer Diagnosis to Palbociclib Initiation [Median (Full Range); unit: Months] — The date of palbociclib treatment initiation was the study baseline. Here, time from initial breast cancer diagnosis to palbociclib initiation was reported. Population: Here, number anaylzed signifies participants evaluable for this baseline measure.
  Months
    number analyzed (Participants) | 541 | 255 | 796
    (all) | 6.0 [0.0 to 397.5] | 27.0 [0.0 to 295.9] | 15.3 [0.0 to 397.5]
Time From Advanced/Metastatic Diagnosis to Palbociclib Initiation [Median (Full Range); unit: Months] — The date of palbociclib treatment initiation was the study baseline. Here, time from advanced/metastatic diagnosis to palbociclib initiation is reported. Population: Here, number anaylzed signifies participants evaluable for this baseline measure.
  Months
    number analyzed (Participants) | 539 | 258 | 797
    (all) | 1.8 [0.0 to 232.6] | 1.4 [0.0 to 128.1] | 1.7 [0.0 to 232.6]

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Rate at Month 6
Description: Progression free rate was defined as percentage of participants who were progression free at defined time point. Progression free was defined as the time from palbociclib combination treatment initiation until the earliest of 1) clinician-documented disease progression while on palbociclib; 2) death; 3) start of a new therapy line after final palbociclib dose if the reason for discontinuation of palbociclib was disease progression; 4) last available follow-up. Disease progression (PD): greater than equal to (>=) 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study, sum must demonstrate absolute increase of at least 5 millimeter (mm) or appearance of 1 or more new lesions. Participants who did not experience a progression event (items 1, 2, 3) were censored at date of last available follow-up. Progression free rate was estimated by Kaplan-Meier analysis.
Time Frame: Month 6 (from the data collected and observed retrospectively for approximately 22 months)
Population: FAS comprised of participants for whom a complete medical record review was conducted. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 573 | 273
Percentage of participants | 93.4 | 91.3

2. Primary Outcome: Progression Free Rate at Month 12
Description: Progression free rate was defined as percentage of participants who were progression free at defined time point. Progression free was defined as the time from palbociclib combination treatment initiation until the earliest of 1) clinician-documented disease progression while on palbociclib; 2) death; 3) start of a new therapy line after final palbociclib dose if the reason for discontinuation of palbociclib was disease progression; 4) last available follow-up. PD: >=20% increase in sum of diameters of target lesions, taking as reference smallest sum on study, sum must demonstrate absolute increase of at least 5 mm or appearance of 1 or more new lesions. Participants who did not experience a progression event (items 1, 2, 3) were censored at date of last available follow-up. Progression free rate was estimated by Kaplan-Meier analysis.
Time Frame: Month 12 (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 573 | 273
Percentage of participants | 80.9 | 76.3

3. Primary Outcome: Progression Free Rate at Month 18
Description: as for outcome 2
Time Frame: Month 18 (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 573 | 273
Percentage of participants | 68.8 | 66.2

4. Primary Outcome: Progression Free Rate at Month 24
Description: as for outcome 2
Time Frame: Month 24 (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 573 | 273
Percentage of participants | 60.9 | 56.1

5. Primary Outcome: Objective Response Rate
Description: Objective response rate was defined as the percentage of participants achieving complete response (CR) or partial response (PR) on palbociclib combination therapy. CR was defined as complete resolution of all visible disease per the treating physicians opinion. PR was defined as partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease.
Time Frame: From date of palbociclib combination treatment initiation to date of CR or PR, up to maximum of 37.4 months (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 572 | 272
Percentage of participants | 69.8 | 67.3

6. Primary Outcome: Percentage of Participants Alive After 1 Year Post Palbociclib Combination Treatment Initiation
Description: Percentage of participants who were alive after 1 year post palbociclib combination treatment initiation were based on the Kaplan-Meier estimate.
Time Frame: 1 year post palbociclib combination treatment initiation (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 557 | 265
Percentage of participants | 95.0 | 96.9

7. Primary Outcome: Percentage of Participants Alive After 2 Years Post Palbociclib Combination Treatment Initiation
Description: Percentage of participants who were alive after 2 years post palbociclib treatment initiation were based on the Kaplan-Meier estimate.
Time Frame: 2 years post palbociclib combination treatment initiation (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 557 | 265
Percentage of participants | 83.0 | 88.8

8. Primary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate was defined as the percentage of participants achieving CR, PR or stable disease (SD) >=24 weeks on palbociclib combination therapy. CR was defined as complete resolution of all visible disease per the treating physicians opinion. PR was defined as partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease. SD was defined as no evidence of complete or partial response, and no progression on palbociclib therapy for 24 weeks or greater. Participants with 12-24 weeks follow up data who remained on palbociclib for the duration of their follow up without evidence of CR or PR or PD were censored.
Time Frame: From date of palbociclib combination treatment initiation to date of PD, up to maximum of 37.4 months (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 572 | 272
Percentage of participants | 94.2 | 95.2

9. Primary Outcome: Percentage of Participants With Stable Disease >=24 Weeks on Palbociclib
Description: SD was defined as no evidence of complete or partial response, and no progression on palbociclib therapy for 24 weeks or greater.
Time Frame: From date of palbociclib combination treatment initiation to date of SD, up to maximum of 37.4 months (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 572 | 272
Percentage of participants | 24.5 | 23.2

10. Primary Outcome: Survival Rate at Month 6
Description: Survival rate was defined as percentage of participants who were not deceased at defined time points. Survival was defined as time from the date of initiation of palbociclib combination therapy to the date of death due to any cause or end of follow-up (if earlier). Survival rate was estimated by Kaplan-Meier analysis.
Time Frame: Month 6 (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 557 | 265
Percentage of participants | 98.9 | 99.6

11. Primary Outcome: Survival Rate at Month 12
Description: as for outcome 10
Time Frame: Month 12 (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 557 | 265
Percentage of participants | 95.0 | 96.9

12. Primary Outcome: Survival Rate at Month 18
Description: as for outcome 10
Time Frame: Month 18 (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 557 | 265
Percentage of participants | 87.7 | 91.2

13. Primary Outcome: Survival Rate at Month 24
Description: as for outcome 10
Time Frame: Month 24 (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 557 | 265
Percentage of participants | 83.0 | 88.8

14. Primary Outcome: Time From Palbociclib Initiation to Initial Response Recorded
Description: CR was defined as complete resolution of all visible disease per the treating physicians opinion. PR was defined as partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease. PD: >=20% increase in sum of diameters of target lesions, taking as reference smallest sum on study, sum must demonstrate absolute increase of at least 5 mm or appearance of 1 or more new lesions. SD was defined as no evidence of complete or partial response, and no progression on palbociclib therapy for 24 weeks or greater.
Time Frame: From date of palbociclib initiation to date of first documented CR, PR, SD or PD, up to maximum of 37.4 months (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 505 | 237
Months | 3.2 [0.1 to 27.6] | 3.0 [0.0 to 15.8]

15. Primary Outcome: Time From Palbociclib Initiation to Complete Response
Description: CR was defined as complete resolution of all visible disease per the treating physicians opinion.
Time Frame: From date of palbociclib initiation to date of first documented CR, up to maximum of 37.4 months (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 51 | 72
Months | 4.5 [1.0 to 27.6] | 4.0 [0.5 to 16.3]

16. Primary Outcome: Time From Palbociclib Initiation to Partial Response
Description: PR was defined as partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease.
Time Frame: From date of palbociclib initiation to date of first documented PR, up to maximum of 37.4 months (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 315 | 95
Months | 3.2 [0.1 to 19.4] | 3.2 [0.0 to 10.3]

17. Primary Outcome: Follow-up Time Since Palbociclib Initiation
Time Frame: From date of palbociclib combination treatment initiation until end of follow-up, maximum of 37.4 months (from the data collected and observed retrospectively for approximately 22 months)
Population: FAS comprised of participants for whom a complete medical record review was conducted.
Measure: Median (Full Range); unit: Months
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 574 | 273
Months | 12.7 [6.0 to 37.4] | 10.7 [3.0 to 36.0]

18. Primary Outcome: Number of Participants With Supportive Therapies
Description: Number of participants who received supportive therapies during palbociclib treatment were reported.
Time Frame: as for outcome 17
Population: FAS comprised of participants for whom a complete medical record review was conducted. Participants could receive more than one supportive treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 574 | 273
Participants
  Bisphosphonates | 246 | 88
  Non-steroidal anti-inflammatory drugs | 232 | 88
  Opioid extended release | 100 | 79
  Anti-emetics | 53 | 19
  Anti-anxiety drugs | 85 | 34
  Anti-depressants | 43 | 56
  Opioid immediate release | 47 | 20
  Other supportive care | 35 | 56
  Antibiotics | 51 | 19
  Nutritional support | 46 | 68
  Granulocyte colony stimulating factors | 24 | 7
  Antifungals | 9 | 2
  Unknown | 2 | 2
  Red blood cell transfusion | 37 | 11
  Pruritus/rash treatments | 5 | 1
  Erythropoietin stimulating agents | 3 | 2
  Platelet transfusions | 7 | 4
  Antivirals | 1 | 15

19. Primary Outcome: Duration of Ongoing Palbociclib Treatment
Time Frame: Up to maximum of 37.4 months (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 391 | 142
Months | 11.2 [6.0 to 37.4] | 8.5 [3.0 to 31.5]

20. Primary Outcome: Duration of Discontinued Palbociclib Treatment
Time Frame: Up to maximum of 37.4 months (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 183 | 131
Months | 8.0 [0.3 to 27.5] | 5.0 [1.0 to 25.1]

21. Primary Outcome: Number of Participants According to Therapies Received Post Palbociclib Treatment
Description: Number of participants who received therapies post palbociclib treatment were reported.
Time Frame: Up to maximum of 37.4 months (from the data collected and observed retrospectively for approximately 22 months)
Population: FAS comprised of participants for whom a complete medical record review was conducted.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 574 | 273
Participants
  Palbociclib / IBRANCE and Fulvestrant/FASLODEX | 0 | 34
  Palbociclib/IBRANCE andFulvestrant/FASLODEX,Exemestane/AROMASIN,Methotrexate | 0 | 2
  Palbociclib/IBRANCE andFulvestrant/ FASLODEX,Letrozole/FEMARA | 0 | 1
  Palbociclib/IBRANCE andFulvestrant/FASLODEX,Methotrexate | 0 | 7
  Palbociclib/IBRANCE andFulvestrant/ FASLODEX,Tamoxifen/NOLVADEX,Methotrexate | 0 | 1
  Palbociclib/IBRANCE andLetrozole/ FEMARA | 4 | 0
  Anastrozole/ARIMIDEX | 2 | 1
  Capecitabine/XELODA | 15 | 15
  Docetaxel/TAXOTERE | 6 | 1
  Docetaxel/TAXOTERE,Capecitabine / XELODA | 3 | 1
  Doxorubicin/ADRIAMYCIN | 1 | 0
  Doxorubicin/ADRIAMYCIN,Cyclophosphamide/CYTOXAN | 1 | 0
  Everolimus/AFINITOR andExemestane/AROMASIN | 11 | 7
  Exemestane/AROMASIN | 6 | 3
  Fulvestrant/FASLODEX | 16 | 1
  Gemcitabine/GEMZAR | 4 | 0
  Nab Paclitaxel/ABRAXANE | 1 | 2
  Other | 0 | 1
  Paclitaxel/TAXOL | 13 | 4
  Paclitaxel/TAXOL,Capecitabine / XELODA | 1 | 0
  Paclitaxel/TAXOL,Doxorubicin/ ADRIAMYCIN,Cyclophosphamide/CYTOXAN | 1 | 0
  Paclitaxel/TAXOL,Gemcitabine/ GEMZAR | 1 | 0
  Palbociclib/IBRANCE and Anastrozole /ARIMIDEX,Methotrexate | 0 | 1
  Palbociclib/ IBRANCE and Exemestane / AROMASIN,Capecitabine/XELODA | 1 | 0
  Palbociclib / IBRANCE and Fulvestrant/FASLODEX,Ixabepilone /IXEMPRA | 0 | 1
  Ribociclib / KISQALI and Exemestane / AROMASIN,Epirubicin /PHARMORUBICIN | 1 | 0
  Tamoxifen / NOLVADEX | 3 | 1
  Tamoxifen / NOLVADEX,Doxorubicin / ADRIAMYCIN | 0 | 1
  Toremifene / FARESTON | 1 | 0
  No treatment | 482 | 188

22. Primary Outcome: Time From Palbociclib Initiation to First Dose Reduction
Time Frame: Up to a maximum of 37.4 months (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 103 | 24
Months | 3.7 [0.7 to 21.8] | 3.4 [0.6 to 13.3]

23. Primary Outcome: Duration of Dose Interruption
Time Frame: Up to a maximum of 37.4 months (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 12 | 1
Days | 14.0 [7.0 to 106.0] | 21.0 [21.0 to 21.0]

24. Primary Outcome: Duration of Cycle Delays
Time Frame: Up to a maximum of 37.4 months (from the data collected and observed retrospectively for approximately 22 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
Number analyzed (Participants) | 2 | 4
Days | 24.5 [14.0 to 35.0] | 21.0 [7.0 to 31.0]

ADVERSE EVENTS:
Time Frame: All-cause mortality data was collected up to 37.4 months post palbociclib combination treatment initiation (from the data recorded during 22 months approximately of retrospective observation period). Data for non-serious adverse events and serious adverse events (SAEs) were not collected and evaluated during the study; hence timeframe is not applicable for non-SAEs and SAEs
Description: Due to non-interventional nature of the study, data for non-SAEs and SAEs were not collected. The study was a retrospective study of existing medical records. There was no collection of adverse events in the study, so there is no report of adverse events in the results.
Arm/Group | Palbociclib + Aromatase Inhibitor | Palbociclib + Fulvestrant
All-Cause Mortality (participants affected / at risk) | 54/574 | 15/273
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT05155566/Prot_SAP_000.pdf